CLINICAL TRIAL: NCT05708001
Title: Improvement of Memory in Mild Cognitive Impairment (MCI) Using Transcranial Alternating Current Stimulation (tACS) Guided by EEG and MRI: a Randomized, Sham-controlled, Parallel-arm, Double-blind Study
Brief Title: Improvement of Memory in Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucie Bréchet (Other)
Responsible Party: Sponsor-Investigator, Lucie Bréchet, Sponsor-Investigator, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-D0055
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: autobiographical memory (ABM); memory and cognition; transcranial alternating current stimulation (tACS); high-density electroencephalography (hdEEG)
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial alternating current stimulation (tACS) (Experimental): The randomized, sham-controlled, parallel-arm, double-blind clinical trial will include 4 weeks of daily, home-based stimulation sessions. MCI patients will be randomly assigned to the active or sham group.
  Interventions: Device: transcranial alternating current stimulation (tACS)
- neurophysiological (hdEEG) (Experimental): At the baseline and after 4 weeks, MCI patients will be evaluated in the laboratory using hdEEG.
  Interventions: Device: high-density electroencephalography (hdEEG)
- clinical measures (MoCA) (Experimental): At the baseline and after 4 weeks, MCI patients will be evaluated in the laboratory using MoCA.
  Interventions: Diagnostic Test: Montreal Cognitive Assessment (MoCA)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — tACS will be delivered by a battery-driven current stimulator Starstim SS32 (Neuroelectrics) through surface Ag/AgCl electrodes placed into holes of a neoprene cap corresponding to the international 10/20 EEG system. Gel (Parker Lab, Inc.) will be applied to optimize signal conductivity and lower impedance. Two tACS (active and sham) conditions will be applied in randomized order. 40 Hz tACS will be delivered to different brain areas of the memory network. We will employ a multielectrode montage based on electric field modeling using the individual MRI to optimally reach the target areas. The maximum injected current per electrode is 2mA and the overall maximal current is 4mA to generate an average electric field of 0.25 V/m.
  Arms: Transcranial alternating current stimulation (tACS)
Device: high-density electroencephalography (hdEEG) — EEG will be recorded with a 257-channel EEG system. An EEG net is applied at once on the head with evenly spaced sensors that provide full scalp coverage, including the cheek. The net contains Ag/Ag-Cl electrodes that are interconnected by thin rubber bands and contain small sponges soaked with saline water that touch the participant's scalp surface directly. Net application takes about 10 min to derive to impedances of <30 kOhms. EEG is recorded with 1 kHz and band-pass filtered between DC-200 Hz. Vertex electrode Cz is used as an acquisition reference.
  Arms: neurophysiological (hdEEG)
Diagnostic Test: Montreal Cognitive Assessment (MoCA) — Clinical Evaluation and Cognitive Assessment - to characterize the level of dementia and changes in cognitive status measured at the baseline and after 4 weeks of gamma/sham tACS intervention, and in a follow-up 3 months after the stimulation using MoCA.
  Arms: clinical measures (MoCA)

SUMMARY:
The Clinical Trial will systematically examine the feasibility of remote, caregiver-led tACS for older adults with memory deficits and evaluate whether repeated tACS leads to sustained improvement of neuronal activity and memory functions.

DETAILED DESCRIPTION:
The proposed investigation will systematically examine the feasibility and efficacy of remote, caregiver-led tACS for older adults with memory decline. This study will provide data to support the safety and effectiveness of home-based tACS in this population and will lead to future research to increase access to tACS as a part of memory decline prevention and treatment for older adults.

ELIGIBILITY:
Inclusion Criteria:

Mild Cognitive Impairment (MCI) patients

* age ≥ 55 years old
* clinical diagnosis of mild cognitive impairment (MCI) based on a comprehensive clinical assessment and standard neuropsychological examination including tests of language, visuospatial thinking, executive functions, and memory
* confirmation of diagnosis will be made by Prof. Paul Unschuld, the study MD, based on a participant's cognitive evaluation and history
* understanding of the informed consent
* able and willing to comply with all study requirements
* informed consent form was signed
* women of childbearing potential (WOCBP) must perform a pregnancy test during screening

Caregiver

* minimum 21 years of age
* self-reported computer/tablet proficiency
* willingness to learn how to use tACS
* availability during the study period to administer tACS to the participant
* informed consent form was signed
* women of childbearing potential (WOCBP) must perform a pregnancy test during screening

Exclusion Criteria:

Mild Cognitive Impairment (MCI) patients

* age < 55 years old
* any current diagnosis of a psychiatric disorder (e.g., schizophrenia, bipolar disorder, depressive disorder)
* other than MCI, any history of other progressive or genetic neurologic disorder (e.g., Parkinson's disease, multiple sclerosis, tubular sclerosis) or acquired neurological disease (e.g., stroke, traumatic brain injury, tumor), including intracranial lesions
* history of head trauma resulting in prolonged loss of consciousness
* current history of poorly controlled headaches including chronic medication for migraine prevention
* history of fainting spells of unknown or undetermined etiology that might constitute seizures
* history of seizures, diagnosis of epilepsy
* any unstable medical condition or chronic uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* contraindication for undergoing MRI or receiving tACS
* any metal in the brain or skull (excluding dental fillings) or elsewhere in the body unless cleared by the responsible covering MD (e.g., MRI compatible joint replacement)
* any skin problems, such as dermatitis, psoriasis, or eczema
* any electrically, magnetically, or mechanically activated implanted devices such as a pacemaker, intracranial electrodes, implanted defibrillators, medication pumps, nerve stimulators, vascular clips, or any other prosthesis in the brain
* any serious life-threatening disease such as congestive heart failure, pulmonary obstructive chronic disease, or active neoplasia
* pregnant women
* adults lacking capacity for consent

Caregiver

* insufficient understanding of study procedures
* poor eyesight, severe arthritis in the hands, pain, deformity or other condition that interferes with successful administration of tACS

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
cognitive status measured by Montreal Cognitive Assessment (MoCA) | baseline, after 4 weeks
  The primary objective is to characterize cognitive status at baseline and after 4 weeks of the home-based stimulation intervention.

SECONDARY OUTCOMES:
modulation of gamma activity assessed with high-density EEG | baseline, after 4 weeks,
  The secondary objective is to assess with hdEEG any changes in gamma power at baseline and after 4 weeks of the home-based stimulation intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Bréchet, PhD, Principal Investigator — University of Geneva (UNIGE); Paul G Unschuld, PhD, Study Chair — Geneva University Hospitals (HUG)
Locations (1):
- University of Geneva, Campus Biotech, Geneva, Switzerland

REFERENCES:
- [Background] Brechet L, Brunet D, Birot G, Gruetter R, Michel CM, Jorge J. Capturing the spatiotemporal dynamics of self-generated, task-initiated thoughts with EEG and fMRI. Neuroimage. 2019 Jul 1;194:82-92. doi: 10.1016/j.neuroimage.2019.03.029. Epub 2019 Mar 19. PMID 30902640
- [Background] Brechet L, Michel CM, Schacter DL, Pascual-Leone A. Improving autobiographical memory in Alzheimer's disease by transcranial alternating current stimulation. Curr Opin Behav Sci. 2021 Aug;40:64-71. doi: 10.1016/j.cobeha.2021.01.003. Epub 2021 Feb 14. PMID 34485630
- [Background] Brechet L, Yu W, Biagi MC, Ruffini G, Gagnon M, Manor B, Pascual-Leone A. Patient-Tailored, Home-Based Non-invasive Brain Stimulation for Memory Deficits in Dementia Due to Alzheimer's Disease. Front Neurol. 2021 May 20;12:598135. doi: 10.3389/fneur.2021.598135. eCollection 2021. PMID 34093384
- [Background] Benussi A, Cantoni V, Grassi M, Brechet L, Michel CM, Datta A, Thomas C, Gazzina S, Cotelli MS, Bianchi M, Premi E, Gadola Y, Cotelli M, Pengo M, Perrone F, Scolaro M, Archetti S, Solje E, Padovani A, Pascual-Leone A, Borroni B. Increasing Brain Gamma Activity Improves Episodic Memory and Restores Cholinergic Dysfunction in Alzheimer's Disease. Ann Neurol. 2022 Aug;92(2):322-334. doi: 10.1002/ana.26411. Epub 2022 Jun 6. PMID 35607946